CLINICAL TRIAL: NCT05735509
Title: Comparison of Scanning With and Without Rubber Dam for Overlay Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Miguel Roig Cayón, Professor, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REST-ECL-2023-01
Record Dates: First submitted 2023-01-29; First posted 2023-02-21 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Crowns
MeSH Terms: interventions — Rubber Dams

STUDY DESIGN:
Intervention Model Description: Tooth to be restored are randomly assigned to on of two groups. In one impressions are taken before placing the rubber dam and in the second impressions are taken after placing the rubber dam.
Who Masked: Investigator
Masking Description: The caree provider takes two impressions and the investigator selects one of them for crown manufacturing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Before rubber dam (Active Comparator): Impression taken before rubber dam placement is used for crown manufacturing
  Interventions: Device: Rubber dam
- After rubber dam (Experimental): Impression taken after rubber dam placement is used for crown manufacturing
  Interventions: Device: Rubber dam

INTERVENTIONS:
Device: Rubber dam — Intraoral impressions can be taken with rubber dam in place. The care provider will take two impressions, one with the rubber dam in place and one without. The investigator will randomly chose one of the two impressions for crown manufacturing, and the crown will be delivered by the care provider blindly

SUMMARY:
The use of rubber dam when performing adhesive restorations improves the quality of the treatment. The widespread use of this type of restorations makes it increasingly necessary to use this type of isolation of the operative field. At the same time, the use of CAD/CAM systems in dentistry has recently become more widespread, which means that chairside systems are being used more and more frequently. Given that in indirect restorations it is necessary to place the rubber dam at the time of cementation, it has been proposed to take optical impressions of the preparation with the rubber dam already in place. For this it is necessary to have previous records that are cut out and rescanned. Since there are authors who have described that rescanning can cause defects in the meshes, in this work we try to compare both types of scanning in a specific type of restorations, the overlays. For this purpose, scans of the tooth preparation with and without rubber dam are taken, and a random decision is made on the basis of which scan the restoration is made. Then it is taken to the mouth and the marginal fit, contact points and occlusion of the restoration are evaluated. The results of the group made from the scan without dam are compared with those of the group made from the scan with dam. The two scans of each case are also compared to evaluate the differences.

DETAILED DESCRIPTION:
1. Introduction: The use of rubber dam in restorative dentistry is important in order to improve the quality of restorations. The incorporation of CAD/CAD systems has led to an increase in the use of chairside techniques. In this work we intend to study in vivo to what extent the optical impressions obtained with rubber dam are equivalent to those taken without rubber dam. For better standardization, overlay restorations are studied.
2. Aims: To compare overlay restorations obtained from a scan with rubber dam placed versus restorations of the same type obtained with a scan without rubber dam.
3. Material and methods:

   (a) Number of patients to be treated: 30. b) Number of visits per patient: 1 c) Brief description of the different techniques used in the study, authorized and validated in the literature (3-5 lines). The use of overlay restorations is widely validated in the literature. In the digital era, rubber dam and non-rubber dam impressions are described in the literature and are used interchangeably. As there is no clinical evidence that both techniques have the same clinical efficacy, we decided to perform this in vivo comparison study.

   d) Benefits and harms for the patient of participating in the study (3-5 lines). Participation in the study does not involve any harm to the patient. It is all performed in the same working time, with identical materials and identical clinical technique. It does not bring any particular benefit to the patient. It is explained to the patient that his/her participation contributes to the improvement of scientific knowledge without physical, economic or material cost.

   e) Alternative treatment in case the patient does not wish to participate in the clinical study (3-5 lines). The same treatment is given whether the patient participates or not. The patient is informed that an overlay is required, the possible complications of this treatment are explained to him/her, and if he/she accepts, he/she is asked if he/she would object to participate in the study. Participation involves consenting to the analysis of the scans and the final evaluation of the restoration.

   f) Treatment to be carried out in the event of complications arising in the patient, once the clinical study has begun (3-5 lines). The clinical study is performed in a single visit and is independent of possible complications of the restoration or the tooth.

   g) Material necessary to carry out the study (3-5 lines). Intraoral anesthesia, milling burs, a Primescan intraoral scanner, rubber dam, W8A clamp, two-step adhesive, 5% hydrofluoric acid, silane, clamp holder, dam drill, glycerin are required. No specific material is required for the study with respect to that required for a patient who does not wish to participate in the study.
4. Evaluation of experimental and statistical results (3 lines). The sample was calculated by means of G power 3 version 3.1.9 software, 80% power and alpha=0.05. A sample of 30 was determined. The Kappa index will be used to evaluate the concordance between the two evaluators, interpreting the results with the Landis and Koch concordance table. Pearson's test will be used to evaluate the fit, occlusal contacts, interproximal contact points and choice of the best impression.

ELIGIBILITY:
Inclusion Criteria:

* Need of an overlay restoration

Exclusion Criteria:

* No need of overlay restoration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-03-05 (Actual); Study Completion 2023-03-05 (Actual)

PRIMARY OUTCOMES:
overall result of final crown | One day
  The final crown is judged by the care provider. A 10 cm Visual analogue scale (VAS) is used. 0 (unacceptable) is placed in left end, and 10 (perfect) is placed in the right end.
Marginal fit of final crown | One day
  Marginal fit will be assessed with an exploratory probe under x3.50 magnification, observing the existence of marginal fit in mesial, distal, buccal, and lingual surfaces. The probe used will be a #23/6 explorer which measures 0.22 mm at 1 mm from the tip. A score of 0 (no perception of the gap when probing), 1 (tip of the probe slightly entered the gap), and 2 (the tip clearly entered the gap) will be used
Contact points fit | One day
  Interproximal contact points will be assessed with waxed dental floss. A score of 0 (incorrect contact point), 1 (correct contact point) will be used
Occlusal adjustment | One day
  Occlusal contacts will be verified with Bausch Arti-Check Micro-Thin 40μ articulating paper and Arti-Fol Metallic Shimstock-Film 12 μ. A score of 0 (no occlusal contacts), 1 (correct occlusal contacts) and 2 (too high occlusal contacts) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: José Espona, DDS, Principal Investigator — Universidad Internacional de Catalunya
Locations (1):
- Clinica Universitaria d'Odontologia, Sant Cugat Del Vallés, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
All data will be published

REFERENCES:
- [Background] Henarejos-Domingo V, Clavijo V, Blasi A, Madeira S, Roig M. Digital scanning under rubber dam: An innovative method for making definitive impressions in fixed prosthodontics. J Esthet Restor Dent. 2021 Oct;33(7):976-981. doi: 10.1111/jerd.12787. Epub 2021 May 18. PMID 34008328
- [Derived] Espona J, Roig E, Ali A, Vidal C, Garcia-Font M, Roig M, Figueras O. Optical impressions assessment for overlay restorations with rubber dam: A clinical trial. J Dent. 2024 Apr;143:104825. doi: 10.1016/j.jdent.2023.104825. Epub 2023 Dec 28. PMID 38157974